CLINICAL TRIAL: NCT03584204
Title: Role of Skeletal Muscle Parameters in Imaging Analysis in the Prediction of Outcome in Patients With Liver Cirrhosis
Brief Title: Skeletal Muscle Parameters of Liver Cirrhosis in Non-invasive Imaging and Outcome
Acronym: SLIM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Michael Praktiknjo, Principal Investigator, University Hospital, Bonn
Other Study IDs: SLIM
Record Dates: First submitted 2018-05-08; First posted 2018-07-12 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Liver Cirrhosis
Keywords: sarcopenia; cirrhosis; transjugular intrahepatic portosystemic shunt; TIPS; acute-on-chronic liver failure; ACLF
MeSH Terms: conditions — Liver Cirrhosis; Sarcopenia; Fibrosis; Acute-On-Chronic Liver Failure | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: imaging — computed tomography, magnetic resosnance imaging, ultrasound

SUMMARY:
The principal aim of this study is to analyse L3-SMI (skeletal muscle index) in a cohort of patients with decompensated liver cirrhosis and TIPS (transjugular intrahepatic portosystemic shunt), and compare the prognostic power with TPMT (transverse psoas muscle thickness). Furthermore, the role of myosteatosis, determined in CT by L3-SMI, MRI and ultrasound will be studied.

DETAILED DESCRIPTION:
The principal aim of this study is to analyse L3-SMI (skeletal muscle index) in a cohort of patients with decompensated liver cirrhosis and TIPS (transjugular intrahepatic portosystemic shunt), and compare the prognostic power with TPMT (transverse psoas muscle thickness). Furthermore, the role of myosteatosis, determined in CT by L3-SMI, MRI and ultrasound will be studied.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis of any etiology
* CT scan available

Exclusion Criteria:

* HCC or any malignant disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis of any etiology and CT scan available
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Survival time | up to 60 months
  time of survival

SECONDARY OUTCOMES:
Time to clinical acute decompensations | up to 60 months
  time to occurrence of acute decompensations of liver cirrhosis (readmissions, hepatic encephalopathy, bleeding, ascites, hepatorenal syndrome, infections)
Time to clinical acute-on-chronic liver failure | up to 60 months
  acute-on-chronic liver failure according to EASL-CLIF-C definition (grade 1 (best) to 3 (worst)
Development of sarcopenia | up to 60 months
  Assessment of sarcopenia according to EASL-guideline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Praktiknjo, MD, Principal Investigator — University Hospital, Bonn
Locations (3):
- Germany (2):
  - University Hospital Bonn, Bonn
  - University of Frankfurt, Frankfurt
- Sapienza University of Rome, Roma, Italy

REFERENCES:
- [Derived] Praktiknjo M, Zhou T, Krusken M, Jacob T, Sprinkart AM, Nowak S, Kimmann M, Dold L, Chang J, Jansen C, Strassburg CP, Luetkens J, Weismuller TJ. Myosteatosis independently predicts transplant-free survival in patients with primary sclerosing cholangitis. Dig Liver Dis. 2023 Nov;55(11):1543-1547. doi: 10.1016/j.dld.2023.08.037. Epub 2023 Aug 14. PMID 37586906
- [Derived] Faron A, Abu-Omar J, Chang J, Bohling N, Sprinkart AM, Attenberger U, Rockstroh JK, Luu AM, Jansen C, Strassburg CP, Trebicka J, Luetkens J, Praktiknjo M. Combination of Fat-Free Muscle Index and Total Spontaneous Portosystemic Shunt Area Identifies High-Risk Cirrhosis Patients. Front Med (Lausanne). 2022 Apr 12;9:831005. doi: 10.3389/fmed.2022.831005. eCollection 2022. PMID 35492329
- [Derived] Queck A, Thomas D, Jansen C, Schreiber Y, Ruschenbaum S, Praktiknjo M, Schwarzkopf KM, Mucke MM, Schierwagen R, Uschner FE, Meyer C, Claria J, Zeuzem S, Geisslinger G, Trebicka J, Lange CM. Pathophysiological role of prostanoids in coagulation of the portal venous system in liver cirrhosis. PLoS One. 2019 Oct 23;14(10):e0222840. doi: 10.1371/journal.pone.0222840. eCollection 2019. PMID 31644538
- [Derived] Praktiknjo M, Clees C, Pigliacelli A, Fischer S, Jansen C, Lehmann J, Pohlmann A, Lattanzi B, Krabbe VK, Strassburg CP, Arroyo V, Merli M, Meyer C, Trebicka J. Sarcopenia Is Associated With Development of Acute-on-Chronic Liver Failure in Decompensated Liver Cirrhosis Receiving Transjugular Intrahepatic Portosystemic Shunt. Clin Transl Gastroenterol. 2019 Apr;10(4):e00025. doi: 10.14309/ctg.0000000000000025. PMID 30939488